CLINICAL TRIAL: NCT00175500
Title: A Randomized Multi-Centre Controlled Trial of Large Diameter (36/40 mm) Versus Conventional Diameter (32 mm) Femoral Heads for the Prevention of Post Revision Arthroplasty Dislocation
Brief Title: Comparison of Conventional and Large Diameter Femoral Heads for the Prevention of Hip Dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C02-0530
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Hip Dislocation
Keywords: Post-Arthroplasty Hip Dislocation
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Large Diameter Femoral Head

SUMMARY:
About ten percent of revision hip replacements will dislocate. Although dislocation is not a life-threatening problem, it is stressful and costly and requires hospitalization to treat. Subjects who have repeated dislocations live with the constant fear of another dislocation. The purpose of this study is to test the effectiveness of a large ball prosthesis in preventing post-surgical dislocation. A large diameter ball has greater freedom of movement before it impinges; therefore, theoretically, it should not dislocate as easily.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients will be those undergoing revision hip arthroplasty, either first revision or subsequent re-revision.
2. Revision must require replacement of both the acetabular component and femoral component, except when revising femur only with well-fixed Trilogy socket.
3. The acetabular component must have a minimum outer diameter of 50 mm.
4. The femoral component inserted should be a Zimmer Versys™ beaded full-coated stem or Zimmer ZMR™ stem or collarless polished taper (CPT™)
5. Patients must be able to reply to questionnaires in either French or English.

Exclusion Criteria:

1. Patients who are undergoing revision for recurrent dislocation.
2. Revision of the acetabulum requiring structural allograft or reconstruction ring.
3. Revision of the acetabulum requiring the use of cemented all-polyethylene cups.
4. Revision of the acetabulum using a liner cemented into an existing metal shell.
5. Intra-operative decision to use a constrained liner.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To compare the difference in dislocation rate between those receiving a large ball (36/40 mm femoral head) versus those receiving a 32 mm femoral head in patients who undergo revision hip arthroplasty | at two years

SECONDARY OUTCOMES:
To compare polyethylene wear in the two groups
To compare the difference in functional and quality of life measures in the two groups | at 3, 12 and 24 months post surgery
To compare radiographic findings in the two groups
To estimate the rate of re-revision in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Donald Garbuz, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada